CLINICAL TRIAL: NCT00164242
Title: Treatment of Tardive Dyskinesia With Galantamine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Caroff, Stanley N., M.D. (Individual)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 00347; 00347
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Tardive Dyskinesia
Keywords: Tardive dyskinesia; Galantamine; Cholinesterase inhibitors
MeSH Terms: conditions — Tardive Dyskinesia | interventions — Galantamine

INTERVENTIONS:
Drug: Galantamine

SUMMARY:
Tardive dyskinesia (TD), a form of movement disorder, remains a problem for some patients who received antipsychotic medications. Increasing evidence suggests that TD may result from antipsychotic-induced dysfunction in striatal cholinergic neurons. To test whether cholinesterase inhibitors compensate for diminished cholinergic activity underlying TD, we conducted a 30-week randomized, double-blind, placebo-controlled crossover study of galantamine in 36 patients with TD.

DETAILED DESCRIPTION:
BACKGROUND: Tardive dyskinesia (TD) is an infrequent but important complication of treatment with antipsychotic medications. Although newer antipsychotics may be less likely to cause TD, it still occurs among some mentally ill patients previously treated with typical antipsychotics. Although usually mild, TD may be more troublesome in some patients. There is no proven curative or suppressive treatment that is effective in all patients. Suppressive treatment with cholinergic agents derives from a hypothesized balance between dopaminergic and cholinergic neurotransmission in the extrapyramidal system. Although previous trials of cholinergic precursors have been unsuccessful in treating TD, their effect on central cholinergic neurotransmission remains uncertain in view of evidence of damage to striatal cholinergic neurons in patients with TD. In contrast, the recent development of cholinesterase inhibitors that are effective in modifying the central cholinergic deficit in Alzheimer's disease, prompted us to investigate the therapeutic effect of galantamine in patients with TD.

RESEARCH OBJECTIVES: We propose to complete a randomized, double-blind, placebo-controlled crossover trial in 36 patients to test; (1) whether galantamine is pharmacologically active in suppressing TD; (2) whether doses of 8-24 mg/day are sufficient for improvement; (3) whether there are any significant side effects in these patients.

METHODS: Thirty-six patients with abnormal involuntary movements meeting research criteria for TD, who are on stable doses of psychotropic medications, will be randomized to receive galantamine alternating with placebo in addition to their standard medications. After 2 baseline measurements, each patient will undergo 12-week treatment periods of galantamine and placebo with a 4-week washout period between treatments. Patients will be evaluated every 2 weeks throughout the study, using standardized rating scales for TD (AIMS) and other extrapyramidal side effects (SIMPSON, BARNES. During the active treatment period, patients will receive galantamine 4 mg BID for 4 weeks followed by 8 mg BID for 4 weeks, and 12 mg BID for an additional 4 weeks. Placebo-galantamine differences will be examined by repeated measures analysis of covariance for a two-period crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of tardive dyskinesia lasting at least 3 months
* Treatment with antipsychotic drugs at least for 3 months
* 18 years old or older

Exclusion Criteria:

* Significant active medical illness
* Allergy to galantamine
* Pregnancy
* Drug or alcohol dependence
* Necessary use of anticholinergics or vitamin E

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2002-01; Study Completion 2004-10

PRIMARY OUTCOMES:
Change in Abnormal Involuntary Movement scale at 3 months.

SECONDARY OUTCOMES:
Change in Simpson-Angus and Barnes Akathisia scales at 3 moths.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley N Caroff, MD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center
Locations (1):
- Philadelphia VA Medical Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Caroff SN, Campbell EC, Havey J, Sullivan KA, Mann SC, Gallop R. Treatment of tardive dyskinesia with donepezil: a pilot study. J Clin Psychiatry. 2001 Oct;62(10):772-5. doi: 10.4088/jcp.v62n1004. PMID 11816865
- [Derived] Caroff SN, Walker P, Campbell C, Lorry A, Petro C, Lynch K, Gallop R. Treatment of tardive dyskinesia with galantamine: a randomized controlled crossover trial. J Clin Psychiatry. 2007 Mar;68(3):410-5. doi: 10.4088/jcp.v68n0309. PMID 17388711